CLINICAL TRIAL: NCT05408585
Title: Minimum Effective Concentration (MEC90) for Supra-inguinal Fascia Iliaca Block Performed Under Ultrasound Guidance in Arthroscopic Knee Surgery
Brief Title: MEC90 for Supra-inguinal Fascia Iliaca Block Performed Under Ultrasound Guidance in Arthroscopic Knee Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsun University (Other)
Collaborators: Samsun Education and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MEC90
Record Dates: First submitted 2022-05-30; First posted 2022-06-07 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: As suggested by Durham et al and described by Dixon, study randomization will be performed using the biased-coin design up-down sequential method.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: All blocks will be performed by the same experienced anesthetist to ensure block quality and homogeneity. The anesthetist applying the block will not take part in the patient follow-up, the independent assistant following the patient will be blinded to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SIFIB with concentration "A" (Active Comparator): The patients were placed in a supine position, and their skin was disinfected and draped. A linear ultrasonography probe was positioned parasagittally and slightly medially on the anterior superior iliac spine. The sartorius, iliacus, internal oblique muscles and deep circumflex iliac artery were visualized. A 80-mm peripheral nerve block needle was advanced, using the in-plane technique, from cranial to caudal until the tip was positioned between the internal oblique and iliacus muscles. Suprainguinal fascia iliaca block will be performed with concentration "A".
  Interventions: Other: Regional Anesthesia Techniques
- SIFIB with concentration "B" (Active Comparator): The patients were placed in a supine position, and their skin was disinfected and draped. A linear ultrasonography probe was positioned parasagittally and slightly medially on the anterior superior iliac spine. The sartorius, iliacus, internal oblique muscles and deep circumflex iliac artery were visualized. A 80-mm peripheral nerve block needle was advanced, using the in-plane technique, from cranial to caudal until the tip was positioned between the internal oblique and iliacus muscles.Suprainguinal fascia iliaca block performed with concentration "B"
  Interventions: Other: Regional Anesthesia Techniques

INTERVENTIONS:
Other: Regional Anesthesia Techniques — Fascial Plane Blocks

SUMMARY:
In this study, the minimum effective concentration required for supra-inguinal fascia iliaca block applied in patients undergoing arthroscopic knee surgery is aimed. The same volume will be used in all of the block applications in the study, and the local anesthetic concentration used will be determined by increasing or decreasing according to the success of the previous block. The primary goal of the study is block success.

DETAILED DESCRIPTION:
For patients included in the study, 40 mL of local anesthetic will be used for SIFIB. The local anesthetic concentration will be randomized using the biased-coin design up-down sequential method, as suggested by Durham et al. and described by Dixon.

The primer outcome of this study is block success. Also, the incidence of motor block formation in the quadriceps muscle (to be defined as paresis or paralysis in knee extension), the amount of tramadol needed in 24 hours, opioid-related side effects (postoperative nausea/vomiting, itching), length of hospital stay and complications that may develop related to the block will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing arthroscopic knee surgery under spinal anesthesia will be included in the study.

Exclusion Criteria:

* Conditions where regional anesthesia is contraindicated (coagulopathy, infection..)
* Patients who underwent general anesthesia for the surgical procedure
* Patients who do not want to be included in the study by not signing the voluntary consent form.
* Patients with advanced dementia, orientation-cooperation problems
* History of allergy to local anesthetic drugs
* Infection status at the injection site

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
Block Success | at 6, 12, 24 hours
  Block success will be evaluated on the post-operative period in the antrior and lateral of thigh using pinprick test.

SECONDARY OUTCOMES:
Tramadol Consumption | 24 hours
  Tramadol Consumption in 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: SERKAN TULGAR, M.D., Study Director — CLINICAL CHIEF
Locations (1):
- Samsun University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dixon WJ. Staircase bioassay: the up-and-down method. Neurosci Biobehav Rev. 1991 Spring;15(1):47-50. doi: 10.1016/s0149-7634(05)80090-9. PMID 2052197
- [Result] Durham SD, Flournoy N, Rosenberger WF. A random walk rule for phase I clinical trials. Biometrics. 1997 Jun;53(2):745-60. PMID 9192462